CLINICAL TRIAL: NCT00306358
Title: Plasma Holotranscobalamin as Compared to Plasma Cobalamins for Assessment of Vitamin B12 Absorption. Optimisation of a Non-Radioactive Vitamin B12 Absorption Test (CobaSorb)
Brief Title: Plasma Holotranscobalamin as Compared to Plasma Cobalamins for Assessment of Vitamin B12 Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20050067
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Vitamin B12 Absorption
Keywords: absorption test; cobalamin; holotranscobalamin; vitamin B12
MeSH Terms: interventions — Vitamin B 12

INTERVENTIONS:
Drug: Vitamin B12 (Cyanocobalamin)

SUMMARY:
In the present study the design of the vitamin B12 absorption test, CobaSorb, is further optimised. We investigate which test - measurement of holotranscobalamin or cobalamins - could be used for reflection of vitamin B12 absorption. Furthermore, we prolong the duration of vitamin B12 administration in order to determine the final duration of the vitamin B12 absorption test CobaSorb.

Seventy-eight healthy individuals (age 21-81 years) are treated with three oral doses of 9 microgram cyanocobalamin per day for five successive days. Non-fasting blood samples are collected on day 1-5 before administration of the first dose of vitamin B12 and on day 8. Cobalamins and holotranscobalamin are measured on day 1-5 and 8. The performance of the vitamin B12 absorption test will be evaluated in individuals with borderline or low levels of holotranscobalamin or cobalamins (below the 75% percentiles) using a change larger than 2CV(day to day) of holotranscobalamin (22%) and cobalamins (12%) to indicate a change caused by absorption of the administered vitamin B12.

DETAILED DESCRIPTION:
In the present study the design of the vitamin B12 absorption test, CobaSorb, is further optimised. We investigate which test - measurement of holotranscobalamin or cobalamins - could be used for reflection of vitamin B12 absorption. Furthermore, we prolong the duration of vitamin B12 administration in order to determine the final duration of the vitamin B12 absorption test CobaSorb.

Seventy-eight healthy individuals (age 21-81 years) are treated with three oral doses of 9 microgram cyanocobalamin per day for five successive days. Non-fasting blood samples are collected on day 1-5 before administration of the first dose of vitamin B12 and on day 8. Cobalamins and holotranscobalamin are measured on day 1-5 and 8. The performance of the vitamin B12 absorption test will be evaluated in individuals with borderline or low levels of holotranscobalamin or cobalamins (below the 75% percentiles) using a change larger than 2CV(day to day) of holotranscobalamin (22%) and cobalamins (12%) to indicate a change caused by absorption of the administered vitamin B12.

ELIGIBILITY:
Inclusion Criteria:

Above 18 years North european origin Read and understand Danish

Exclusion Criteria:

Vitamin B12 treatment within the past 5 years Use of vitamin pills containing >1 microgram vitamin B12 with in the past 3 weeks Infectious disease Pregnancy Lactation Giving birth within the past 9 months Use of hormones Known systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Start 2005-05; Study Completion 2005-10

PRIMARY OUTCOMES:
Changes in plasma holotranscobalamin after intake of vitamin B12

SECONDARY OUTCOMES:
Changes in plasma cobalamins, plasma methylmalonic acid and plasma homocysteine after intake of vitamin B12.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, Cand Med PhD, Principal Investigator — Dept. of Clinical Biochemistry, Skejby Sygehus, 8000 Aarhus, Denmark
Locations (1):
- Aarhus Sygehus, Aarhus, Denmark